CLINICAL TRIAL: NCT00121251
Title: A Phase I/II Trial of BAY 43-9006 Plus Gemcitabine and Capecitabine in the Treatment of Patients With Advanced Renal Cell Carcinoma
Brief Title: Sorafenib, Gemcitabine, and Capecitabine in Treating Patients With Unresectable and/or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00108; NCI-2009-00108 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000434851; 0501007709 (Other: Montefiore Medical Center - Moses Campus); 6981 (Other: CTEP); N01CM62204 (NIH); P30CA013330 (NIH)
Record Dates: First submitted 2005-07-19; First posted 2005-07-21 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Recurrent Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v7; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Capecitabine; Gemcitabine; Sorafenib

ARMS (1):
- Sorafenib + Gemcitabine + Capecitabine (Experimental): Patients receive sorafenib* PO BID on days 1-21, gemcitabine IV over 30 minutes on days 1 and 8, and capecitabine PO BID on days 1-14. Treatment repeats every 21 days for at least 3 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: Capecitabine; Drug: Gemcitabine Hydrochloride; Drug: Sorafenib Tosylate

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This phase I/II trial is studying the side effects and best dose of sorafenib, gemcitabine, and capecitabine and to see how well they work in treating patients with unresectable and/or metastatic kidney cancer. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with gemcitabine and capecitabine may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of sorafenib administered in combination with gemictabine and capecitabine in patients with advanced renal cell carcinoma.

II. Determine the objective response rate for sorafenib in combination with gemictabine and capecitabine in patients with advanced renal cell carcinoma.

III. Determine the duration of overall survival and progression free survival in these patients.

OUTLINE: This is a multicenter, non-randomized, phase I dose-escalation study followed by a phase II study.

PHASE I: Patients receive sorafenib* orally (PO) twice daily (BID) on days 1-21, gemcitabine intravenously (IV) over 30 minutes on days 1 and 8, and capecitabine PO BID on days 1-14. Treatment repeats every 21 days for at least 3 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of sorafenib, gemcitabine, and capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 6 patients are treated at the MTD.

Note: *Patients who complete at least 3 courses of treatment with objective response or stable disease but are deemed poor candidates for continued chemotherapy may continue treatment with sorafenib

PHASE II: Patients receive sorafenib 200mg orally twice a day on days 1-21, gemcitabine 750 mg/m2 intravenously on days 1 & 8, and capecitabine 415 mg/m2 orally twice a day on days 1-14 of each 21 day cycle, as in phase I at the MTD determined in phase I.

After completion of study treatment patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed renal cell carcinoma that is unresectable and/or metastatic; patients with collecting duct carcinoma, oncocytomas, or transitional cell carcinoma are not eligible; patients with sarcomatoid renal cell carcinoma are eligible, but those with pure sarcomas are not; histologic documentation of metastatic disease is not required; clinical confirmation, but not pathologic staging, of metastatic disease is required
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Patients may have received one prior immunotherapy based regimen (i.e. interleukin-2 or interferon alpha) ending >= 4 weeks prior to enrollment
* Patients may have received up to 2 prior regimens containing mitogen-activated protein kinases (MAPK), vascular endothelial growth factor (VEGF) pathway inhibitors (e.g. sunitinib or bevacizumab) and/or mammalian target of rapamycin (mTOR) inhibitor (e.g. temsirolimus) ending >= 4 weeks prior to enrollment
* Life expectancy of more than 3 months
* Eastern Cooperative Oncology Group (ECOG) =< 2 OR Karnofsky >= 60%
* Leukocytes >= 3000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelet count >= 100,000/uL
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x IULN
* Creatinine =< 1.5 x IULN OR creatinine clearance >= 60 mL/min/1.73m^2 for patients with creatinine levels above institutional normal
* The effects of sorafenib on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because raf kinase inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not have received prior chemotherapy; if patients have had prior definitive or other surgery, prior radiation therapy, they must have fully recovered from the effects of therapy with at least 4 weeks recovery time; for patients who have had a surgical biopsy only, they must have simply recovered
* Patients may not be receiving any other investigational agents
* Patients with known active brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; previously treated brain metastases are allowed if they show no evidence of progression on CT or magnetic resonance imaging (MRI) at least 8 weeks after completion of surgery and/or radiotherapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib, gemcitabine and capecitabine
* No concurrent megestrol is permitted; no megestrol therapy within 4 weeks prior to protocol treatment is allowed; no concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, phenobarbitol or carbamazepine), rifampin, or St. John's wort
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary disease including asthma, chronic bronchitis, emphysema with requirements for chronic oxygen use or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because sorafenib is a kinase inhibitor agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sorafenib, breastfeeding should be discontinued if the mother is treated with sorafenib; the potential risks may apply to other agents used in this study
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with sorafenib, gemcitabine, or capecitabine administered during the study; appropriate studies will be undertaken in patients receiving combination ant-retroviral therapy when indicated
* Any swallowing dysfunction leading to difficulty taking the investigational therapy or capecitabine
* Prior treatment with sorafenib
* Patients with any history or evidence of a bleeding diathesis
* Patients on therapeutic anticoagulation with coumarins (e.g. warfarin); prophylactic coumarin-based anticoagulation (i.e. low dose warfarin) for venous or arterial access devices is allowed provided that the requirements for prothrombin time (PT), international normalization ratio (INR) and/or partial thromboplastin time (PTT) are met; prophylactic or therapeutic low molecular weight heparin is allowed; patients with known brain metastases are excluded (even if treated and stable) if they are also on therapeutic doses of anticoagulation
* Patients with known dihydropyrimidine dehydrogenase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-06-03 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, Principal Investigator — Montefiore Medical Center - Moses Campus
Locations (4):
- United States (4):
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to enrollment in June 2005 and closed to enrollment September 2011. Patients were recruited from the inpatient and outpatient clinics at Weill Cornell Medical Center, Columbia University Medical Center, North Shore Hospital, New York University Hospital, Montefiore Medical Center, Mount Sinai Medical Center and others
Period: Overall Study
Arm/Group | Sorafenib + Gemcitabine + Capecitabine
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib + Gemcitabine + Capecitabine
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 62 [41 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Status [Count of Participants; unit: Participants]
  0 Normal Activity | 4
  1 Symptoms, but ambulatory. Restricted in strenuous activities | 10
  2 Capable of all self-care but unable to carry out any work activities. In bed <50% of the time | 3
Histology [Count of Participants; unit: Participants]
  Papillary | 6
  Clear Cell | 8
  Sarcomatoid | 1
  Chromophobe | 1
  Unclassified | 1
Site of Metastasis [Count of Participants; unit: Participants]
  Lung/Pleura | 14
  Lymph Node | 9
  Liver | 3
  Bone | 1
  Other Viscera | 10
  2 or more sites | 15
Previous Treatment [Count of Participants; unit: Participants]
  Nephrectomy | 15
  Cytokines | 1
  Sunitinib | 1
MSK Classification [Count of Participants; unit: Participants]
  Favorable | 5
  Intermediate | 9
  Poor | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response for BAY 43-9006 in Combination With Gemcitabine and Capecitabine Evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR
Time Frame: Up to 9 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib + Gemcitabine + Capecitabine
Number analyzed (Participants) | 17
Participants | 5

2. Secondary Outcome: Median Number of Months of Progression Free Survival (PFS)
Description: PFS will be measured from the time of the patient's initial best response (PR or CR) until documented progression.
Time Frame: From the time of the patient's initial best response (PR or CR) until documented progression, assessed up to 9 years
Measure: Median (Full Range); unit: Months
Arm/Group | Sorafenib + Gemcitabine + Capecitabine
Number analyzed (Participants) | 17
Months | 5 [3 to 17]

3. Secondary Outcome: Number of Participants Who Survived (Overall Survival)
Description: Overall survival (OS) is defined as the time from start of treatment to death from any cause.
Time Frame: Up to 9 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib + Gemcitabine + Capecitabine
Number analyzed (Participants) | 17
Participants | 6

ADVERSE EVENTS:
Time Frame: Up to 9 years
Arm/Group | Sorafenib + Gemcitabine + Capecitabine
All-Cause Mortality (participants affected / at risk) | 11/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 5/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib + Gemcitabine + Capecitabine (N=17)
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-05-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT00121251/Prot_SAP_000.pdf